CLINICAL TRIAL: NCT01200186
Title: Non-interventional Study on Oral Contraception Not Containing Ethinylestradiol (EE) to Assess Continuation Rates and Satisfaction
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15217; QL0901 (Other: Company Internal)
Record Dates: First submitted 2010-08-13; First posted 2010-09-13 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Contraceptives, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027)
- Group 2
  Interventions: Drug: Progestin Only Pills

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027) — At the discretion of the attending physician
  Groups: Group 1
Drug: Progestin Only Pills — At the discretion of the attending physician
  Groups: Group 2

SUMMARY:
Prospective, non-interventional, multi-center study. Each subject will be followed for up to twelve months during the treatment with oral hormonal contraceptives(Qlaira ® or a Progestin Only Pill). For each subject demographic data and medical history will be documented at Visit 1: (Baseline). Bleeding profile, subjective assessment of study treatment (satisfaction and wellbeing) and adverse events including unintended pregnancies will be documented at Visit 2 (Month 3-5) and Visit 3 (Month 6-12). Data audit/monitoring will be done.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-50 years
* Women who used ethinylestradiol containing oral contraceptives for at least the three preceding months before the study
* Women who decided to start Qlaira® or a Progestin Only Pill. The prescription of the hormonal contraceptive is made at the discretion of the attending physician and has to be documented

Exclusion Criteria:

* Contraindications and warnings of the respective Summary of Product Characteristics (Qlaira® or Progestin Only Pill)
* Women who are breast-feeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women in gynecological practice
Sampling Method: Non-Probability Sample
Enrollment: 3258 (Actual)
Dates: Start 2010-10; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be time-to-event for discontinuation due to bleeding irregularities. | up to 12 Months

SECONDARY OUTCOMES:
Time to event for discontinuation due to reasons other than bleeding irregularities | Month 3-5
Time to event for discontinuation due to reasons other than bleeding irregularities | Month 6-12
Number of intracyclic bleeding | Month 3-5
Number of intracyclic bleeding | Month 6-12
Number of heavy and/or prolonged bleeding | Month 3-5
Number of heavy and/or prolonged bleeding | Month 6-12
Number of unintended pregnancies | Month 3-5
Number of unintended pregnancies | Month 6-12
Discontinuation rate for the following reasons: Occasional absent or persistent absent withdrawal bleeding , intracyclic bleeding, heavy and/or prolonged bleeding, other medical reasons, non-medical reasons | Month 3-5
Discontinuation rate for the following reasons: Occasional absent or persistent absent withdrawal bleeding , intracyclic bleeding, heavy and/or prolonged bleeding, other medical reasons, non-medical reasons | Month 6-12
Global assessment of well-being and satisfaction | Month 3-5
Global assessment of well-being and satisfaction | Month 6-12
Adverse events (AEs) at any time point, whether or not related to the therapy or reference therapy | up to 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Many Locations, Czechia
- Many Locations, France
- Many Locations, Germany
- Many Locations, Greece
- Many Locations, Hungary
- Many Locations, Israel
- Many Locations, Italy
- Many Locations, Russia
- Many Locations, Slovakia
- Many Locations, Sweden
- Many Locations, United Kingdom